CLINICAL TRIAL: NCT05680857
Title: The Efficacy and Safety of Products Containing Marine Collagen Peptide and Coenzyme Q10 for Skin Rejuvenation in Malaysian Women
Brief Title: Efficacy and Safety of Products Containing Marine Collagen Peptide and Coenzyme Q10 for Skin Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UMRAMREC005-22
Record Dates: First submitted 2022-12-27; First posted 2023-01-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo group will receive a product in sachet form that doesn't have marine collagen peptide and Coenzyme Q10.
  Interventions: Other: Placebo
- Product containing marine collagen peptide and Coenzyme Q10. (Experimental): This group will receive the product containing marine collagen peptide from the fish origin and Coenzyme Q10 in sachet form.
  Interventions: Other: Product containing marine collagen peptide and Coenzyme Q10.

INTERVENTIONS:
Other: Placebo — Product doesn't have active ingredients i.e. marine collagen peptide and Coenzyme Q10.
  Arms: Placebo
Other: Product containing marine collagen peptide and Coenzyme Q10. — Product containing marine collagen peptide and Coenzyme Q10.
  Arms: Product containing marine collagen peptide and Coenzyme Q10.

SUMMARY:
This is a placebo-controlled study conducted to investigates the safety and efficacy of products containing marine collagen peptide and CoQ10 in enhancing skin rejuvenation of Malaysian women. The study duration is 28 days and the skin assessment will be carried out at baseline, Day 14 and Day 28.The main questions it aims to answer are:

1. The effect of product on skin hydration of women in Malaysia.
2. The effect of product on skin elasticity of women in Malaysia.
3. The effect of product on skin wrinkle of women in Malaysia.
4. The skin brightening effect of product on Malaysian women.
5. To observe any adverse effect occurrence with the consumption of the product.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizen
* Women aged 35 - 45 years old
* Willing to participate

Exclusion Criteria:

* Women with skin diseases or any underlying diseases.
* Pregnant, breastfeeding women or planned pregnancy during the study period
* Allergy to collagen or other ingredients that may be found in the product.
* Women who had any cosmetic procedures such as botox, laser and light treatment, facial surgery, and any procedures that may improve skin hydration, elasticity, wrinkles, and brightening of skin four weeks before the study.
* Women who took any dietary supplements, functional foods, or medicines that could have the same or similar effects as the product evaluated in this study in the past three months.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in skin hydration from baseline and at Day 14 and Day 28 after consumption of a product. | Baseline, Day 14 and Day 28
  Skin hydration will be assessed using JANUS III skin analyzer and comparison will be made with placebo group.
Changes in skin elasticity from baseline and at Day 14 and Day 28 after consumption of a product. | Baseline, Day 14 and Day 28
  Skin elasticity will be assessed using JANUS III skin analyzer comparison will be made with placebo group.
Changes in skin wrinkles from baseline and at Day 14 and Day 28 after consumption of a product. | Baseline, Day 14 and Day 28
  Skin wrinkles will be assessed using JANUS III skin analyzer comparison will be made with placebo group.
Changes in skin tone from baseline and at Day 14 and Day 28 after consumption of a product. | Baseline, Day 14 and Day 28
  Skin hydration will be assessed using JANUS III skin analyzer comparison will be made with placebo group.
Adverse effect after consumption of product containing marine collagen peptide and coenzyme Q10. | 28 Days
  Based on adverse effect occurrence on participants that occur during study period (28 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No